CLINICAL TRIAL: NCT02861508
Title: Impact of Immediate Point-of-Care Ultrasound on Patients With Cardiopulmonary Symptoms in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1605017729
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Chest Pain; Dyspnea; Syncope; Hypotension
Keywords: Ultrasonography
MeSH Terms: conditions — Chest Pain; Dyspnea; Syncope; Hypotension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Usual care as determined by treating team. Ultrasound may still be part of the workup per the treating team's discretion.
  Interventions: Other: Usual care
- Early POCUS (Experimental): Point-of-care ultrasound protocol will involve cardiac views (for pericardial effusion, left ventricular function, left and right ventricular equality, aortic root dilation, and inferior vena cava status), lung views (for pneumothorax, signs of alveolar interstitial syndrome), abdominal views for free fluid, and a view of the abdominal aorta for aneurysm.
  Interventions: Other: Point-of-care ultrasound

INTERVENTIONS:
Other: Point-of-care ultrasound
  Arms: Early POCUS
Other: Usual care
  Arms: Usual care

SUMMARY:
The purpose of the proposed research is to examine whether incorporating point-of-care ultrasound (POCUS) early in diagnostic work-up of cardiopulmonary complaints will affect diagnosis, time to condition-specific intervention, and ultimately patient outcomes compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Chief complaint of chest pain, dyspnea (either sudden onset or increased severity of chronic dyspnea), syncope, or hypotension (systolic blood pressure <100 or shock index [heart rate divided by systolic blood pressure] >1)

Exclusion Criteria:

* <18 years old
* Prisoner or ward of the state
* Trauma
* High acuity requiring treatment in resuscitation room
* Obvious cause of symptoms (e.g. acute GI bleed causing hypotension)
* Any form of "do not resuscitate" (DNR) order
* Roomed in hall of emergency department (location not amenable to ultrasound protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Time to appropriate intervention | Within 30 days of presentation
  Based on final diagnosis as determined by final review of the patient's overall visit in the medical record, it will be determined what the appropriate intervention(s) that the patient should have received. Subsequently, the amount of time that elapsed (minutes) between time the patient was roomed in the emergency department (ED) and time to when they received the intervention will be collected. All these time points are readily available in the electronic medical record in the patient care timeline. This outcome will help determine whether early POCUS affects how quickly patients receive appropriate intervention.

SECONDARY OUTCOMES:
Diagnostic accuracy | Within 30 days of presentation
  The treating team in the ED will be asked for their diagnostic impression of the patient's chief complaint at several points during the patient's time in the ED. These points will be (1) after the primary provider's initial assessment, (2) at time of disposition, and (3) if they are in the early POCUS group, after the POCUS findings are relayed to them. They will select their single most likely diagnosis each time, which will be compared against a final diagnosis as determined by final review of the patient's overall visit in the medical record (as this study's gold standard for diagnosis). This outcome will examine how often (percentage-wise) the treating team's diagnosis matches the final diagnosis as well as if early POCUS has any impact on helping physicians reach the correct diagnosis.
Diagnostic certainty | Within 2 days of presentation
  Similar to the outcome of diagnostic accuracy, the treating team in the ED will concomitantly be asked how certain they feel about their diagnosis on a five-point scale. The presence of any changes in certainty (i.e. proportion of patients for whom certainty changed) as well as how much change (e.g. increased certainty by 2 points) will be assessed. This outcome will determine if early POCUS affects physicians' certainty of diagnosis.
Time to disposition | Within 2 days of presentation
  This will be measured as amount of time (in minutes) that elapse between the time patient is roomed in the ED to time the treating team determines patient disposition. These timestamps are available in the medical record under the patient care timeline. This outcome will examine if early POCUS affects the time it takes for the treatment team to achieve a disposition plan for the patient.
Total length of stay | Within 30 days of presentation
  This will be measured as time (in days) between the patient's date of presentation and date of discharge. This outcome will examine if early POCUS affects the amount of time that patients stay in the hospital.
30-day in-hospital mortality | Within 30 days of presentation
  Patients will be followed in their medical record for up to 30 days after their initial presentation to assess for in-hospital mortality rate. This outcome will examine if early POCUS leads to any significant difference in patient mortality rate compared to usual care.
Duration of POCUS | Within 2 days of presentation
  For the early POCUS group, this will be measured as the amount of time (in minutes) between the time the ultrasound is started and the time the last image is captured. All images/video clips acquired by the ultrasound machine have a timestamp. A blank image will be captured at the start of the exam for the initial timestamp. This outcome will examine how time-consuming our POCUS exam is and provides a sense of how disruptive the introduction of POCUS might be if it were implemented routinely.

OTHER OUTCOMES:
Return visits with missed diagnosis | Within 30 days of presentation
  The patient's medical record will be followed for 30 days after initial presentation for the presence of any repeat visits with the healthcare system for a similar chief complaint. If so, that repeat visit will be reviewed for the presence of a different diagnosis than that established at the original visit, which would suggest that the correct diagnosis had been missed at that time. It will then be determined what the percentage of patients is with such visits out of all patients in the study. This outcome will examine if POCUS helps with picking up diagnoses that might be missed otherwise.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Moore, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
No specific plans for now but would be open to sharing anonymized data.